CLINICAL TRIAL: NCT05114681
Title: Oral Care in Stroke Patients: An Observational Study of a Tertiary Care Center
Brief Title: Oral Health Care in Stroke Patients in Tertiary Care Hospital
Status: Completed | Type: Observational
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Responsible Party: Principal Investigator, Muhammad Hassan, Registrar Neurology, Shaheed Zulfiqar Ali Bhutto Medical University
Other Study IDs: Dental care in stroke
Record Dates: First submitted 2021-10-29; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: Gingivitis; Periodontitis; Dental Hygiene
MeSH Terms: conditions — Gingivitis; Periodontitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment of Oral care as per patient personal choice — We just inquire from patients or attendants about products used, the timing for oral care.

SUMMARY:
To investigate oral care provision in stroke care settings in Pakistan. Stroke can have adverse effects on oral care and health. Little is known about current oral care practices in stroke care settings.

DETAILED DESCRIPTION:
For a variety of related reasons, stroke can adversely affect oral care. Physical impairment, coordination, sensory or cognitive deficits may accompany a stroke and can impact on independent oral care. Post-stroke alterations in facial muscle mass or movement and sensory problems may result in poorly controlled dentures.

Dysphagia can contribute to oral care concerns in a number of ways. Oral intake of fluids may be restricted to reduce the risk of aspiration pneumonia, which in turn can contribute to xerostomia. Nutritional supplements, often prescribed, are high in sugar and may predispose to caries. Furthermore, because of swallowing impairment, pharmacological interventions are often administered in syrup consistency, which is sugar-based, and may also predispose to caries. Reduced swallowing ability causes ineffective clearance of bacteria and debris from the mouth leading to caries and infection.

Some pharmacological interventions in stroke care are known to have oral side effects. Oxygen therapy frequently administered in acute stroke management is known to cause mucosal drying and blistering. The absence of normal chewing patterns as a result of pain, physical or sensory impairment can also reduce salivary function. Xerostomia also causes pain, taste disturbance, chewing, and swallowing difficulties.

Speech and denture retention is also affected by inadequate saliva. This, in turn, increases plaque formation, predisposes to opportunistic oral infections, periodontal disease, and caries, conditions which place the individual at greater risk of pain, tooth loss and tooth substance loss. Chronic periodontal infection is currently being tentatively linked with the incidence of the stroke itself, while others have demonstrated a relationship with other systemic diseases including pneumonia and cardiovascular disease.

Healthcare-led oral care is a complex intervention and comprises a number of elements. These include assessment, accessing further assistance as required, and the use of appropriate equipment and cleaning methods. Knowledge is also required to assess and apply oral care at an individual level.

ELIGIBILITY:
Inclusion Criteria:

* Patient with diagnosed case of stroke
* Both gender will be included.

Exclusion Criteria:

* Patients with a known case of bleeding diathesis.
* patient not willing to participate
* patient with known head and neck cancer and oral pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Stroke
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Assessment of Dental Hygiene | baseline
  assessment of dental hygiene will be done with ROAG scale
Dental care tools survey | baseline
  ask about tools for dental care in stroke units

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Hassan, MD, Principal Investigator — Shaheed Zulfiqar Ali Bhutto Medical University
Locations (1):
- Shaheed Zulfiqar Ali Bhutto Medical University, Islamabad, Capital, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared at reasonable request.